CLINICAL TRIAL: NCT04334083
Title: Biomarkers Of Job STRess In Emergency Senior Physicians - Detection of Stressful Events
Brief Title: Biomarkes Of Job STRess In Emergency Senior Physicians - Detection of Stressful Events
Acronym: JOBSTRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RBHP 2019 DUTHEIL 2; 2019-A02961-56 (Other: 2019-A02961-56)
Record Dates: First submitted 2020-03-25; First posted 2020-04-06 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Heart Rate Variability
Keywords: Heart rate variability; stress; cortisol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emergency physicians (Experimental): actors during the work
  Interventions: Behavioral: Comparison of biomarkers of stress
- medical externship student (Experimental): spectator during the emergency physician work
  Interventions: Behavioral: Comparison of biomarkers of stress

INTERVENTIONS:
Behavioral: Comparison of biomarkers of stress — Emergency will be followed during a night shift and the rest day et during a day shift and the rest day. They will be observed by a medical externship student. We will assess the role of expertise and habituation to stressful emergency situations.

SUMMARY:
Emergency medicine is a unique specialty focusing on a breadth of acute care, on demand . Shift work is also a fundamental component of emergency medicine, and is associated with chronic stress, including stress at work. Consequently, stress may lead to symptoms of mental exhaustion, physical fatigue, detachment from work, and feelings of diminished competence . Emergency physicians (EPs) are exposed to a complex interplay between stress (life-and-death emergencies - a defining characteristic of their job), sleep deprivation, and fatigue due to repeated changes in, and duration of shifts. Work-related exhaustion can lead to various physical and psychological symptoms, and also may be associated with delayed decision-making . The combined effects of stress and fatigue can impact on job performance, often resulting in otherwise preventable medical errors. Moreover, prolonged stress may expose EPs to a higher risk of multiple diseases, predominantly systemic inflammation and coronary heart disease. All these contribute to the premature departure of EPs to other specialties. Furthermore, low HRV has been associated with stress, burnout, and is linked with an increased risk of cardiovascular diseases.

This project proposes to evaluate if life-and-death emergencies or specific situations will induce abrupt changes in HRV among emergency physicians. Moreover, we would like to compare reactions between being an actor (EPs) and being a spectator and assess the role of expertise and habituation to stressful emergency situations.

DETAILED DESCRIPTION:
The JOBSTRESS protocol was designed to provide a better understanding of the association between specific situations (ie: life and death emergencies) and breaks in the variability of the heart rate. Each emergency physician participates in the study two times. A night shift from 6:30 p.m to 8:30 a.m (14 hours) which will be compared with a day shift, as a control, from 8:30 a.m to 6:30 p.m. Emergency physicians will be accompanied by a medical externship student.

Statistical analysis will be performed using Stata software (version 13; Stata-Corp, College Station, Tex., USA). All statistical tests will be bilateral and a p <0.05 will be considered significant. Qualitative variables will be described in terms of numbers and proportions. Quantitative variables will be described in terms of numbers, average, median, standard deviation, and range. Graphic representations will be complete presentations of results. We process multivariate physiological series (HR, HRV, SC, wrist motion, respiratory rate) in order to build a stress index. For such multivariate physiological series, we first use change point analysis on each univariate series in order to get clusters with constant parameters, then we use classification algorithm on the constant parameters obtained in first step in order to obtain different classes corresponding to different levels of stress. Eventually, we obtain at each time the level of stress and can compare it to the environmental conditions.

ELIGIBILITY:
Inclusion Criteria:

* Emergency physicians from the emergency department of CHU Clermont-Ferrand will be accompanied by a medical externship student.
* Ability to give a written informed consent.

Exclusion Criteria:

* Participant refusal to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
heart rate variability at night work | from 18:30 to 8:30, during the 14 hours of the night shift
  measure of abrupt changes in HRV signals during 14 hours
heart rate variability at day work | from 8:30 to 18:30, during the 10 hours of the day shift
  measure of abrupt changes in HRV signals during 10 hours

SECONDARY OUTCOMES:
Stress | 18:30, baseline of the night shift
  measure of stress using VAS
Fatigue | at 18:30, baseline of the night shift
  measure of Fatigue using VAS
Stress | at 8h30, at the end of the night shift
  measure of stress using VAS
Fatigue | at 8:30, at the end of the night shift
  measure of Fatigue using VAS
Stress | at 8:30, 24 hours after the end of night shift
  measure of stress using VAS
Fatigue | at 8:30, 24 hours after the end of night shift
  measure of Fatigue using VAS
Fatigue | at 18:30, 24 hours after the end of day shift
  measure of Fatigue using VAS
Stress | at 18:30, 24 hours after the end of day shift
  measure of stress using VAS
Stress | at 8:30, baseline of the day shift
  measure of stress using VAS
Fatigue | at 8:30, baseline of the day shift
  measure of Fatigue using VAS
Stress | at 18:30, end of the day shift
  measure of stress using VAS
Fatigue | at 18:30, end of the day shift
  measure of Fatigue using VAS
Saliva biomarkers cortisol | at 18:30, baseline of the night shift
  measure of Cortisol
Saliva biomarkers cortisol | at 8:30, at the end of the night shift
  measure of Cortisol
Saliva biomarkers cortisol | at 8:30, baseline of the day shift
  measure of Cortisol
Saliva biomarkers cortisol | at 18:30, end of the day shift
  measure of Cortisol
Saliva biomarkers DHEAS | at 18:30, baseline of the night shift
  measure of DHEAS
Saliva biomarkers DHEAS | at 8:30, at the end of the night shift
  measure of DHEAS
Saliva biomarkers DHEAS | at 8:30, baseline of the day shift
  measure of DHEAS
Saliva biomarkers DHEAS | at 18:30, end of the day shift
  measure of DHEAS
Saliva biomarkers lgAs | at 18:30, baseline of the night shift
  measure of lgAs
Saliva biomarkers lgAs | at 8:30, at the end of the night shift
  measure of lgAs
Saliva biomarkers lgAs | at 8:30, baseline of the day shift
  measure of lgAs
Saliva biomarkers lgAs | at 18:30, end of the day shift
  measure of lgAs
blood samples full blood count | at 8:30, at the end of the night shift
  measure of full blood count
blood samples full blood count | at 8:30, baseline of the day shift
  measure of full blood count
blood samples HbA1c, | at 8:30, at the end of the night shift
  measure of HbA1c
blood samples HbA1c, | at 8:30, baseline of the day shift
  measure of HbA1c
blood samples HDLc and LDL-cholesterol | at 8:30, at the end of the night shift
  measure of HDLc and LDL-cholesterol
blood samples HDLc and LDL-cholesterol | at 8:30, baseline of the day shift
  measure of HDLc and LDL-cholesterol
blood samples TG | at 8:30, at the end of the night shift
  measure of TG
blood samples TG | at 8:30, baseline of the day shift
  measure of TG
blood samples Cortisol | at 8:30, at the end of the night shift
  measure of Cortisol
blood samples Cortisol | at 8:30, baseline of the day shift
  measure of Cortisol
blood samples DHEAS | at 8:30, at the end of the night shift
  measure of DHEAS
blood samples DHEAS | at 8:30, baseline of the day shift
  measure of DHEAS
blood samples vitamine D | at 8:30, at the end of the night shift
  measure of vitamine D
blood samples vitamine D | at 8:30, baseline of the day shift
  measure of vitamine D
blood samples BDNF | at 8:30, at the end of the night shift
  measure of BDNF
blood samples BDNF | at 8:30, baseline of the day shift
  measure of BDNF
blood samples proinflammatory cytokines | at 8:30, at the end of the night shift
  measure of proinflammatory cytokines
blood samples proinflammatory cytokines | at 8:30, baseline of the day shift
  measure of proinflammatory cytokines
blood samples telomeres lengh | at 8:30, at the end of the night shift
  measure of telomeres lengh
blood samples telomeres lengh | at 8:30, baseline of the day shift
  measure of telomeres lengh
Burnout | day 1
  Burnout is assessed by the Maslach Burn-out Inventory (MBI) composed by 22 items and a 7-point scale ranging from "never" to "every day".
Depression | day 1
  depression is assessed by the Hospital Anxiety and Depression scale (HAD) composed by 7 items and a 4-point scale from "never" to "always".
Anxiety | day 1
  Anxiety is assessed by the the Hospital Anxiety and Depression scale (HAD) composed by 7 items and a 4-point scale from "never" to "always" and by the State-Trait Anxiety Inventory (STAI) composed by two dimensions, state anxiety and trait anxiety, both evaluated with a 20-items questionnaire on a 4-point scale from "never" to "always".
Life satisfaction | day 1
  quality of life is assessed by a brief multidimensional life satisfaction scale (BMLSS)
Lifestyle | day 1
  Assessing factors regarding lifestyle are related to smoking, alcohol, coffee, food intake (questionnaires), and physical activity (Recent Physical Activity Questionnaire).
Life and occupational events | day 1
  Assessing factors regarding death of patients or death of a loved one by questionnaire.
Sick leave | day 1
  assessing sick leave by the number of absence days the previous 6 months using a questionnaire
Clinical measurements height | day 1
  measure of height
Clinical measurements weight | day 1
  measure of weight
diastolic blood pressure | at 18:30, baseline of the night shift
  measure of diastolic blood pressure
systolic blood pressure | at 18:30, baseline of the night shift
  measure of systolic blood pressure
diastolic blood pressure | at 8:30, at the end of the night shift
  measure of diastolic blood pressure
systolic blood pressure | at 8:30, at the end of the night shift
  measure of systolic blood pressure
diastolic blood pressure | at 8:30, baseline of the day shift
  measure of disatolic blood pressure
systolic blood pressure | at 8:30, baseline of the day shift
  measure of systolic blood pressure
diastolic blood pressure | at 18:30, end of day shift
  measure of disatolic blood pressure
systolic blood pressure | at 18:30, end of day shift
  measure of systolic blood pressure
skin conductance | from 18:30 to 8:30, during the 14 hours of night shift
  measure of the skin conductance
skin conductance | from 8:30 to 18:30, during the 10 hours of day shift
  measure of the skin conductance
Genetic factors ACE | at 8:30, end of the night shift
  measure of the polymorphism of angiotensin converting enzyme inhibitors (ACE
Genetic factors ACE | at 8:30, baseline of the day shift
  measure of the polymorphism of angiotensin converting enzyme inhibitors (ACE
Genetic factors (5-HTT) | at 8:30, end of the night shift
  measure of the polymorphism of the serotonin transporter (5-HTT)
Genetic factors (5-HTT) | at 8:30, baseline of the day shift
  measure of the polymorphism of the serotonin transporter (5-HTT)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Dutheil, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France